CLINICAL TRIAL: NCT03262077
Title: Evaluation of Parameters of Tissue Dosimetry in Photodynamic Therapy for the Treatment of Periodontal Disease - Clinical Study
Brief Title: Dose Parameters for Photodynamic Therapy on Periodontal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Collaborators: Sandra Kalil Bussadori (Unknown)
Responsible Party: Principal Investigator, Renato Araujo Prates, PhD., University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: University of Nove de Julho
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Chronic Periodontitis
Keywords: photodynamic therapy; periodontal disease; dosimetry; methylene blue
MeSH Terms: conditions — Chronic Periodontitis; Periodontal Diseases | interventions — Methylene Blue

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- MB 1 min (Experimental): Methylene blue 100 μM photosensitizer was deposited in the periodontal pocket of one incisor and 1 min of pre-irradiation time was adopted to allow the drug to stain the bacterial biofilm. Then the laser emitting wavelength of 660 nm, with power of 100 mW, was applied to the mucosa during 1 min.
  Interventions: Drug: Methylene Blue
- MB 3 min (Experimental): Methylene blue 100 μM photosensitizer was deposited in the periodontal pocket of one incisor and 1 min of pre-irradiation time was adopted to allow the drug to stain the bacterial biofilm. Then the laser emitting wavelength of 660 nm, with power of 100 mW, was applied to the mucosa during 3 min.
  Interventions: Drug: Methylene Blue
- MB 5 min (Experimental): Methylene blue 100 μM photosensitizer was deposited in the periodontal pocket of one incisor and 1 min of pre-irradiation time was adopted to allow the drug to stain the bacterial biofilm. Then the laser emitting wavelength of 660 nm, with power of 100 mW, was applied to the mucosa during 5 min.
  Interventions: Drug: Methylene Blue
- MBS 1 min (Experimental): Methylene blue photosensitizer 100 μM + soap was deposited in the periodontal pocket of one incisor and 1 min of pre-irradiation time was adopted to allow the drug to stain the bacterial biofilm. Then the laser emitting wavelength of 660 nm, with power of 100 mW, was applied to the mucosa during 1 min.
  Interventions: Drug: Methylene Blue Oral Product
- MBS 3 min (Experimental): Methylene blue photosensitizer 100 μM + soap was deposited in the periodontal pocket of one incisor and 1 min of pre-irradiation time was adopted to allow the drug to stain the bacterial biofilm. Then the laser emitting wavelength of 660 nm, with power of 100 mW, was applied to the mucosa during 3 min.
  Interventions: Drug: Methylene Blue Oral Product
- MBS 5 min (Experimental): Methylene blue photosensitizer 100 μM + soap was deposited in the periodontal pocket of one incisor and 1 min of pre-irradiation time was adopted to allow the drug to stain the bacterial biofilm. Then the laser emitting wavelength of 660 nm, with power of 100 mW, was applied to the mucosa during 5 min.
  Interventions: Drug: Methylene Blue Oral Product

INTERVENTIONS:
Drug: Methylene Blue — Irradiation with low-level laser for 1, 3, and 5 min
  Arms: MB 1 min; MB 3 min; MB 5 min
Drug: Methylene Blue Oral Product — Irradiation with low-level laser for 1, 3, and 5 min
  Arms: MBS 1 min; MBS 3 min; MBS 5 min

SUMMARY:
Due to the phenomenon of bacterial resistance, photodynamic therapy (PDT) has been studied as an alternative to the use of antibiotics on the periodontal treatment. However, the studies show several discrepancies between the parameters adopted for PDT, which makes it difficult to compare the results and measure their efficacy. The objective of this research was to investigate the tissue dosimetric parameters used in PDT for the treatment of periodontal disease. In order to achieve this objective, the scattering pattern of light in periodontal tissue, the concentration of methylene blue in the periodontal pockets and the number of viable microorganisms were evaluated. This clinical trial included 30 patients with chronic periodontitis according to the eligibility criteria. The patients were in periodontal treatment at the Dental Clinic at the University of Nove de Julho, where the research was carried out. Three incisors from each patient were selected for the experimental procedures. The pattern of light scattering was observed through intraoral photographs. A laser with emission of radiation with wavelength of 660 nm and 100 mW of power was used. The concentration of the photosensitizer (PS) in the periodontal pockets was evaluated by spectrometer before irradiation. Methylene blue was used as PS at the concentration of 100 μM in two different formulation and vehicles to evaluate the drug dimerization. Then, the procedures of irradiation of the PDT were carried out, with 3 irradiation times of 1, 3 and 5 min. The microbiological evaluation was performed from subgengival biofilms of the periodontal pockets of the experimental sites, before and immediately after the irradiation procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patient with chronic periodontitis;
* The patient should have at least 15 teeth present, with a minimum of 3 incisors with depth of probing greater than 4 mm;
* The patient should be in periodontal treatment at the Dental Clinic of the University of Nove de Julho, where this research was carried out. All patients were treated according to the protocol recommended by the American Academy of Periodontology;
* Minimum age of 18 years.

Exclusion Criteria:

* current smokers or regular smoking 12 months prior to enrollment;
* patients with anemia,
* patients with active cancer;
* pregnant;
* history of antibiotic therapy in the previous six months;
* history of anti-inflammatory therapy in the previous three months;
* patients with clotting disorders;
* patients currently undergoing orthodontic treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-10-11 (Actual); Primary Completion 2017-06-26 (Actual); Study Completion 2017-06-26 (Actual)

PRIMARY OUTCOMES:
Bacterial reduction | 48 hours after the laser irradiation procedure.
  Count of Colony Forming Units